CLINICAL TRIAL: NCT03993509
Title: Examining the Mechanisms of Anxiety Regulation Using a Novel, Sham-controlled, fMRI-guided rTMS Protocol and a Translational Laboratory Model of Anxiety
Brief Title: Effect of rTMS on Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: 833320
Record Dates: First submitted 2019-06-18; First posted 2019-06-20 (Actual); Results first posted 2025-01-23 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Anxiety; Fear; Anxiety and Fear
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Aims 1 and 2 will be tested using a between-subjects design where 1 group of healthy volunteers will receive 4-day courses of active and sham 1 Hz stimulation to the right dlPFC, while the other group will receive 4-day courses of active and sham 10 Hz stimulation to the right dlPFC. Aim 1, will test the effects of this stimulation on anxiety during the NPU threat task. Aim 2, will test the effects of this stimulation on anxiety-related working memory (WM) deficits using the Sternberg WM paradigm. Aim 3 will be tested using a within-subjects design where this same group of subjects will receive single-pulse active and sham stimulation to the right dlPFC during the Neutral, Predictable, and Unpredictable (NPU) threat task while in the MRI scanner. BOLD activity to the TMS pulses will be the primary outcome measure.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Both the subject and the TMS operator will be blinded as to the study condition (active vs. sham)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- 1 Hz Arm (Experimental): Subjects will receive a continuous train of 1 Hz stimulation until all 3000 pulses are delivered. Consistent with the 10 Hz condition, TMS will occur during the Sternberg WM paradigm.
  Interventions: Device: rTMS to the right dlPFC
- 10 Hz Arm (Experimental): Subjects will receive 75, 4 second trains at 10 Hz, separated by a 36 second ITI. Stimulation will occur while subjects are doing the Sternberg WM paradigm. The timing of the Sternberg task will be jittered so that each rTMS train will be administered during the maintenance interval of a WM trial.
  Interventions: Device: rTMS to the right dlPFC

INTERVENTIONS:
Device: rTMS to the right dlPFC — A Magventure MagPro 100X stimulator with a B65 active/placebo figure-8 coil will be used. The TMS coil will be placed on the head over the target. rTMS intensity will be 100% of the motor threshold (MT), adjusted for field strength difference at motor cortex and target cortex using the individual E-field model. Subjects will receive 3000 pulses/session.

SUMMARY:
Given the overall lack of treatment adherence/efficacy, side effects of drugs, and the substantial burden of anxiety disorders on the individual and on the national healthcare system, there is a critical need for mechanistic research into the CNS mechanisms that underlie these disorders. Accordingly, the objective of this grant is to use noninvasive neuromodulation to causally identify the key neural mechanisms that mediate the cognitive symptoms of anxiety. This project is relevant to public health because it has the potential to lead to novel repetitive transcranial magnetic stimulation treatments for pathological anxiety.

DETAILED DESCRIPTION:
Although extensive research has explored the involvement of subcortical structures in arousal, arousal symptoms are only one facet of the symptom profile shared across anxiety disorders. Much less is known about the cognitive symptoms (i.e. difficulty concentrating) experienced by anxiety patients. Accordingly, there is a critical need for mechanistic research into the CNS mechanisms that mediate the cognitive symptoms experienced by anxiety patients. Without such research, treatment development for these disorders will continue to make slow progress. The objective of this application is to determine the key neural mechanisms that mediate the cognitive symptoms of anxiety. The central hypothesis is that the right dorsolateral prefrontal cortex (dlPFC) regulates emotion through top-down inhibition of emotion-related regions. The approach will be to use repetitive transcranial magnetic stimulation (rTMS) to study the effect of right dlPFC activity on objective and subjective measures of induced anxiety, anxiety-related working memory deficits (WM), and TMS-evoked blood oxygenation-level dependent (BOLD) responses during simultaneous TMS/fMRI (i.e. target engagement). The rationale for this approach is that by experimentally manipulating right dlPFC activity using rTMS, this research will be able to causally demonstrate involvement of this region in anxiety regulation, which could translate to future targeted rTMS treatments for anxiety. The first aim will be to determine the effect of a 1-week course of rTMS treatment (1 Hz vs. 10 Hz; right dlPFC target) on anxiety using the threat of unpredictable shock paradigm. The second aim will be to determine the effect of a 1-week course of rTMS treatment (1 Hz vs. 10 Hz; right dlPFC target) on anxiety-related WM-deficits using the Sternberg WM paradigm during threat of shock. The third aim will be to demonstrate target engagement by measuring BOLD responses evoked by TMS pulses to the right dlPFC during threat of shock. The work is innovative because it will combine advanced neuromodulatory techniques (fMRI guidance, electric-field modelling, neuronavigation, active-sham control) with a translational threat of shock paradigm. PUBLIC HEALTH RELEVANCE: Once completed, this research should yield direct evidence for a causal role of the right dlPFC in anxiety regulation, complete with evidence of target engagement, and a novel application to anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 18-50 years old
* Able to give their consent
* Right-handed

Exclusion Criteria:

* Non-english speaking
* Any significant medical or neurological problems
* Current or past Axis I psychiatric disorder(s), active or history of active suicidal ideation
* Alcohol/drug problems in the past year or lifetime alcohol or drug dependence
* Medications that act on the central nervous system
* History of seizure
* History of epilepsy
* Increased risk of seizure for any reason
* Pregnancy, or positive pregnancy test
* IQ <80
* Any medical condition that increases risk for fMRI or TMS
* Any metal in their body which would make having an MRI scan unsafe
* Any sort of medical implants
* Hearing loss
* Claustrophobia

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2019-10-30 (Actual); Primary Completion 2022-11-23 (Actual); Study Completion 2022-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- cTBS Arm (Active/Sham); cTBS Arm (Sham/Active): Subjects assigned to the cTBS Arm completed both an active and a sham period, separated by a 1-week break. Some subjects received the active period first, while other subjects received the sham period first. The period data below are collapsed across counterbalance.
  Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  cTBS parameters. During each cTBS session, a single 600 pulse cTBS train was delivered during each stimulation session at 100% of RMT. The train consisted of 50 Hz bursts, repeated at intervals of 200 ms (5 Hz) for 40 sec. The active side of the coil was used for these sessions.
- iTBS Arm (Active/Sham); iTBS (Sham/Active): Subjects assigned to the iTBS Arm completed both an active and a sham period, separated by a 1-week break. Some subjects received the active period first, while other subjects received the sham period first. The period data below are collapsed across counterbalance.
  Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  iTBS parameters. During each iTBS session, ten 60-pulse iTBS trains were delivered at 100% of RMT. The trains consisted of 3 50 Hz bursts repeated at intervals of 200 ms (5 Hz) for 2 seconds of stimulation separated by 8 second gaps, for a total of 600 pulses per session.
Period: Active
Arm/Group | cTBS Arm (Active/Sham) | iTBS Arm (Active/Sham) | cTBS Arm (Sham/Active) | iTBS (Sham/Active)
Started | 18 | 17 | 16 | 17
Completed | 15 | 16 | 13 | 14
Not Completed | 3 | 1 | 3 | 3
Period: Sham
Arm/Group | cTBS Arm (Active/Sham) | iTBS Arm (Active/Sham) | cTBS Arm (Sham/Active) | iTBS (Sham/Active)
Started | 15 | 16 | 13 | 14
Completed | 15 | 16 | 13 | 12
Not Completed | 0 | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Population: participants between the ages of 18 and 50 were recruited from the Philadelphia, PA, metropolitan area to take part in this study.
Groups:
- cTBS Arm: Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  cTBS parameters. During each cTBS session, a single 600 pulse cTBS train was delivered during each stimulation session at 100% of RMT. The train consisted of 50 Hz bursts, repeated at intervals of 200 ms (5 Hz) for 40 sec.
- iTBS Arm: Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  iTBS parameters. During each iTBS session, ten 60-pulse iTBS trains were delivered at 100% of RMT. The trains consisted of 3 50 Hz bursts repeated at intervals of 200 ms (5 Hz) for 2 seconds of stimulation separated by 8 second gaps, for a total of 600 pulses per session.
- Total: Total of all reporting groups
Arm/Group | cTBS Arm | iTBS Arm | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.61 (7.04) | 23.75 (4.26) | 25.18 (5.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 18 | 39
  Male | 7 | 10 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 26 | 26 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 6 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 17 | 16 | 33
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 28 | 28 | 56

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Potentiated Startle
Description: Electromyography Facial electromyography (EMG) startle responses were recorded from the left orbicularis oculi muscle at 2000 Hz using a Biopac MP160 unit (Biopac; Goleta, CA) via 15 × 20 mm hydrogel coated vinyl electrodes (Rhythmlink #DECUS10026; Columbia, SC).
  Startle EMG was bandpass filtered from 30 to 300 Hz, rectified, and smoothed using a 20-ms sliding window. Startle responses were scored as the peak (max during the 20 ms to 120 ms post-noise window) - the baseline (50 ms pre-noise window), and converted to t-scores with a mean of 50 and a standard deviation of 10 (tx = [Zx × 10] + 50). Greater t-scores mean larger blinks, which could be associated with greater anxiety, however there is no clinically relevent threshold. Noisy trials (baseline SD > 2x run SD) were excluded, and "no blink" (peak < baseline range) trials were coded as 0. To calculate APS, we subtracted the response during the neutral ITI from the response during the unpredictable ITI.
Time Frame: Pre and 24-hours post stimulation
Measure: Mean (Standard Deviation); unit: T-scores
Groups:
- cTBS Arm (Active/Sham); cTBS Arm (Sham/Active): Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  cTBS parameters. During each cTBS session, a single 600 pulse cTBS train was delivered during each stimulation session at 100% of RMT. The train consisted of 50 Hz bursts, repeated at intervals of 200 ms (5 Hz) for 40 sec.
- iTBS Arm (Active/Sham); iTBS Arm (Sham/Active): Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  iTBS parameters. During each iTBS session, ten 60-pulse iTBS trains were delivered at 100% of RMT. The trains consisted of 3 50 Hz bursts repeated at intervals of 200 ms (5 Hz) for 2 seconds of stimulation separated by 8 second gaps, for a total of 600 pulses per session.
Arm/Group | cTBS Arm (Active/Sham) | iTBS Arm (Active/Sham) | cTBS Arm (Sham/Active) | iTBS Arm (Sham/Active)
Number analyzed (Participants) | 15 | 16 | 13 | 12
T-scores
  active | 4.600026484 (3.690076704) | 3.411297242 (4.494552916) | 3.122643391 (4.286242167) | 4.848463905 (2.77573715)
  sham | 2.098026426 (3.687256948) | 1.347655375 (5.091633437) | 3.063363512 (4.002345814) | 3.551809142 (4.504709597)

2. Primary Outcome: Fear Potentiated Startle
Description: Electromyography Facial electromyography (EMG) startle responses were recorded from the left orbicularis oculi muscle at 2000 Hz using a Biopac MP160 unit (Biopac; Goleta, CA) via 15 × 20 mm hydrogel coated vinyl electrodes (Rhythmlink #DECUS10026; Columbia, SC).
  Startle EMG was bandpass filtered from 30 to 300 Hz, rectified, and smoothed using a 20-ms sliding window. Startle responses were scored as the peak (max during the 20 ms to 120 ms post-noise window) - the baseline (50 ms pre-noise window), and converted to t-scores with a mean of 50 and a standard deviation of 10 (tx = [Zx × 10] + 50). Greater t-scores mean larger blinks, which could be associated with greater fear, however there is no clinically relevent threshold. Noisy trials (baseline SD > 2x run SD) were excluded, and "no blink" (peak < baseline range) trials were coded as 0. To calculate FPS, we subtracted the response during the predictable ITI from the response during the predictable Cue.
Time Frame: Pre and 24 hours post stimulation
Measure: Mean (Standard Error); unit: T-scores
Arm/Group | cTBS Arm (Active/Sham) | iTBS Arm (Active/Sham) | cTBS Arm (Sham/Active) | iTBS Arm (Sham/Active)
Number analyzed (Participants) | 15 | 16 | 13 | 12
T-scores
  active | 7.598819444 (4.007589756) | 6.719283178 (5.508434373) | 6.564791401 (4.771055896) | 5.529855023 (4.175930826)
  sham | 5.61775824 (3.484582125) | 3.016188249 (6.334558956) | 6.651174586 (5.405511643) | 6.496396165 (3.242895129)

3. Primary Outcome: Sternberg WM Accuracy
Description: Sternberg task: On each WM trial, subjects will see a series of 4 letters presented singularly (encoding period) that will be followed by a brief interval where subjects are required to maintain these letters (maintenance period). At the end of the maintenance period, subjects will be prompted to make a response based on the task instructions (response period). The response prompt will consist of a letter and a number. The letter will be chosen from the study series, and the number will correspond to a position in the series. The subjects will indicate whether the position of the letter in the series matches the number.
Time Frame: Pre and 24 hours post stimulation
Measure: Mean (Standard Deviation); unit: percent correct
Groups:
- cTBS (Sham/Active): Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  cTBS parameters. During each cTBS session, a single 600 pulse cTBS train was delivered during each stimulation session at 100% of RMT. The train consisted of 50 Hz bursts, repeated at intervals of 200 ms (5 Hz) for 40 sec.
- iTBS (Sham/Active): Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  iTBS parameters. During each iTBS session, ten 60-pulse iTBS trains were delivered at 100% of RMT. The trains consisted of 3 50 Hz bursts repeated at intervals of 200 ms (5 Hz) for 2 seconds of stimulation separated by 8 second gaps, for a total of 600 pulses per session.
Arm/Group | cTBS Arm (Active/Sham) | iTBS Arm (Active/Sham) | cTBS (Sham/Active) | iTBS (Sham/Active)
Number analyzed (Participants) | 15 | 16 | 13 | 12
percent correct
  active | 80.70887446 (15.81409388) | 86.99776786 (10.46204331) | 84.89010989 (13.40836505) | 87.45039683 (10.42233406)
  sham | 81.38888889 (16.70756441) | 87.85342262 (7.303273682) | 86.76739927 (16.03952935) | 90.35218254 (8.095574634)

4. Primary Outcome: TMS-evoked BOLD Responses
Description: As with Experiment 1, subjects will have Neutral, Predictable, and Unpredictable periods. During the neutral periods, they will be safe from shocks. During the predictable periods, they can receive shocks but only when there is a cue present. During the unpredictable periods, they are at risk for shock during the entire duration of the block. Rather than probing their ongoing anxiety with the startle probes, we replaced the startle probes with single TMS pulses to the right dlPFC. This allowed us to causally examine the effect of right dlPFC activity (induced by the TMS pulse) on the neural activity. BOLD responses are collapsed across regions and conditions to examine right dlPFC BOLD down regulation.
Time Frame: Responses are measured within the TMS/fMRI session in response to each TMS pulse and collapsed across trials. There is no sham condition. This session was typically conducted during the washout period, but varied depending upon participant schedule.
Measure: Mean (Standard Deviation); unit: BOLD signal
Arm/Group | cTBS Arm | iTBS Arm
Number analyzed (Participants) | 22 | 19
BOLD signal | -0.0074 (0.0056) | -0.0063 (0.0072)

ADVERSE EVENTS:
Time Frame: 5 weeks
Description: An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. Intercurrent illnesses or injuries should be regarded as adverse events. Adverse events are classified as serious or non-serious. A serious adverse event is any AE that is: fatal, life-threatening, requires or prolongs hospital stay, results in persistent or significant disability or incapacity a congenital anomaly or birth defect, an important medical event
Groups:
- Active cTBS: Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  cTBS parameters. During each cTBS session, a single 600 pulse cTBS train was delivered during each stimulation session at 100% of RMT. The train consisted of 50 Hz bursts, repeated at intervals of 200 ms (5 Hz) for 40 sec. The active side of the coil was used for these sessions.
- Active iTBS: Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  iTBS parameters. During each iTBS session, ten 60-pulse iTBS trains were delivered at 100% of RMT. The trains consisted of 3 50 Hz bursts repeated at intervals of 200 ms (5 Hz) for 2 seconds of stimulation separated by 8 second gaps, for a total of 600 pulses per session. The active side of the coil was used for these sessions.
- Sham cTBS: Sham stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  cTBS parameters. During each cTBS session, a single 600 pulse cTBS train was delivered during each stimulation session at 100% of RMT. The train consisted of 50 Hz bursts, repeated at intervals of 200 ms (5 Hz) for 40 sec. The sham side of the coil was used for these sessions.
- Sham iTBS: Active stimulation. A Magventure MagPro 100X stimulator with a B65AP (active/placebo) figure-8 coil was used for the cTBS sessions. The active and sham coil sides of the coil were masked and assigned blinded labels (e.g. A = active, B = sham). The label key was maintained by a member of the study staff not directly involved in the collection or analysis of the data. All other study staff were blinded to the label assignments.
  iTBS parameters. During each iTBS session, ten 60-pulse iTBS trains were delivered at 100% of RMT. The trains consisted of 3 50 Hz bursts repeated at intervals of 200 ms (5 Hz) for 2 seconds of stimulation separated by 8 second gaps, for a total of 600 pulses per session. The sham side of the coil was used for these sessions.
Arm/Group | Active cTBS | Active iTBS | Sham cTBS | Sham iTBS
All-Cause Mortality (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34 | 0/34 | 0/34 | 0/34
Other Adverse Events (participants affected / at risk) | 3/34 | 3/34 | 0/34 | 0/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active cTBS (N=34) | Active iTBS (N=34) | Sham cTBS (N=34) | Sham iTBS (N=34)
Mild headache or jaw pain (Product Issues) | 3 (3) | 2 (2) | NA | NA
mild claustrophobia (Product Issues) | 0 (0) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/09/NCT03993509/Prot_SAP_000.pdf